CLINICAL TRIAL: NCT03765996
Title: Effectiveness of Kinesio® Taping on Anastomotic Regions in Patients With Breast Cancer-Related Lymphoedema: A Randomized Controlled Study
Brief Title: Effectiveness of Taping on Anastomotic Regions in Patients With Breast Cancer-Related Lymphoedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ertan Sahinoglu, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2301-GOA
Record Dates: First submitted 2018-12-01; First posted 2018-12-05 (Actual); Results first posted 2020-04-27 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer Lymphedema; Compression Bandages; Manual Lymphatic Drainage
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decongestive Physiotherapy (Active Comparator): This group received Complex Decongestive Physiotherapy.
  Interventions: Other: Decongestive Physiotherapy
- Decongestive Physiotherapy plus taping (Experimental): This group received Complex Decongestive Physiotherapy, and also applying taping to anastomosis regions.
  Interventions: Other: Decongestive Physiotherapy plus taping

INTERVENTIONS:
Other: Decongestive Physiotherapy — This group received CDP, which include MLD, short-stretch bandages, lymph-reducing exercises, and skin care. MLD was applied to the anterior trunk, posterior trunk, and the base of the neck, progressing to the affected limb. Short-stretch bandages were applied in multiple layers after MLD. A low pH skin lotion was applied prior to bandaging and then stockinette was placed on the arm. The fingers and the hand were wrapped in gauze. A layer of cotton was wrapped around the arm. Bandages (6, 8 and/or 10cm) were sequentially applied in a spiral fashion around the limb with the smallest bandage starting at the hand. The most compression was at the most distal points and gradually decreased proximally. Exercises were done by patients to improve mobility and enhance lymphatic flow.
  Arms: Decongestive Physiotherapy
Other: Decongestive Physiotherapy plus taping — This group received CDP as same protocol of active comparator. In addition, Kinesiotaping was applied to anterior and posterior axillo-axillary anastomosis and axillo-inguinal anastomosis. The tape was started on the unaffected side and strips of tape were applied so as to reach the affected side regarding anterior and posterior axillo-axillary anastomosis. For axillo-inguinal anastomosis, the tape was started in the inguinal region of the affected side and strips of tape were applied so that they reached the axillary region.
  Arms: Decongestive Physiotherapy plus taping

SUMMARY:
One of the most common conservative treatments of lymphoedema is Complex Decongestive Physiotherapy (CDP). The bandage is one of the most important components of the treatment process. The multilayer short-stretch bandage is used to maintain volume reduction and prevent lymph backflow caused by compression. However, some patients refuse or postpone treatment or show a lower compliance with compression bandaging.Kinesio® Tex tape (KT) is a new technique for managing lymphoedema in the field of physical and alternative therapy, and it may affect decongestion of lymphatic fluid accumulated under the skin. Some studies which showed that KT was an effective for patients with BCRL, it was applied on both the affected arm and anastomosis. One of these studies also reported that a significant reduction in limb volume in patients who were applied of the tape only to the affected arm. This significant effect could also be seen by applying KT only to the anastomosis. In literature, however, there is no evidence to support this theory. So the aim of this study is to determine the effectiveness of KT which was applied to anastomotic regions along with CDP in the management of BCRL.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had unilateral BCRL and women aged over 18 who were 'significant', 'marked', or 'severe' lymphoedema.

Exclusion Criteria:

* Patients with paralysis on part of the affected arm,
* Patients who had undergone CDP more than once within six months,
* Patients who had an active infection,
* Patients who had a skin disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2015-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gülbin Ergin, PhD, Principal Investigator — European University of Lefke; Didem Karadibak, Prof., Study Director — Dokuz Eylul University; Tuğba Yavuzşen, Prof., Study Director — Dokuz Eylul University
Locations (1):
- Dr. İsmail Atabek Physical Therapy and Rehabilitation Center, Izmir, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled in the study between 2012 and 2014.
Groups:
- Decongestive Physiotherapy Plus Taping: This group received Complex Decongestive Physiotherapy, and also applying taping to anastomosis regions.
  Decongestive Physiotherapy plus taping: This group received CDP as same protocol of active comparator. In addition, taping was applied to anterior and posterior axillo-axillary anastomosis and axillo-inguinal anastomosis. The tape was started on the unaffected side and strips of tape were applied so as to reach the affected side regarding anterior and posterior axillo-axillary anastomosis. For axillo-inguinal anastomosis, the tape was started in the inguinal region of the affected side and strips of tape were applied so that they reached the axillary region.
Period: Overall Study
Arm/Group | Decongestive Physiotherapy | Decongestive Physiotherapy Plus Taping
Started | 18 | 18
Completed | 14 | 18
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decongestive Physiotherapy | Decongestive Physiotherapy Plus Taping | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.42 (7.69) | 58.44 (10.12) | 56.25 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Four patients in control group excluded from the study due to not completed the study
  Participants
    number analyzed (Participants) | 14 | 18 | 32
    Female | 14 | 18 | 32
    Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change of the Limb Volume, (Last Value of the Follow-up - Baseline Value)
Description: Limb size was quantified by using circumferential limb measurements. Measurements were taken with patients in a prone position and the arm abducted at 30°. The circumference was measured every 5cm, starting at the ulnar styloid and continuing 45cm proximally for both limbs. Limb volume was calculated for each segment by using the frustum formula. Frustum formula is a mathematical method for calculating limb volume based on the circumference measures, and this formula gives the result in milliliters. Limb measuring was carried out at the beginning of and after treatment (twenty sessions).
Time Frame: At baseline and at 4 weeks
Measure: Median (Inter-Quartile Range); unit: milliliter
Arm/Group | Decongestive Physiotherapy | Decongestive Physiotherapy Plus Taping
Number analyzed (Participants) | 14 | 18
milliliter | 160.01 [81.50 to 650.56] | 148.28 [52.29 to 552.85]

ADVERSE EVENTS:
Time Frame: up to 4 weeks
Description: Skin deterioration was expected due to bandage or taping, however, any skin allergy or wounds have not occurred in all patients.
Arm/Group | Decongestive Physiotherapy | Decongestive Physiotherapy Plus Taping
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No